CLINICAL TRIAL: NCT04905134
Title: Partnership to Establish a Practice Based Network to Assess for Head and Neck Cancers Using a Low-Cost Portable Flexible Nasopharyngoscope - Optimization Phase
Brief Title: Low-Cost, Portable Flexible Nasopharyngoscope in Head & Neck Cancers in Low Resource Settings - Optimization Phase
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00102912; 1R01DE028555-01A1 (NIH); Protocol Number: 22-136-E (Other: NIDCR)
Record Dates: First submitted 2021-05-24; First posted 2021-05-27 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Head and Neck Cancer; Oral Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Mouth Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Patients evaluated using flexible nasopharyngoscope prototype device (Active Comparator)
  Interventions: Device: Nasopharyngoscope
- Patients evaluated using standard of care nasopharyngoscope (No Intervention)
- Providers using flexible nasopharyngoscope prototype device (Active Comparator)
  Interventions: Device: Nasopharyngoscope

INTERVENTIONS:
Device: Nasopharyngoscope — Low-cost, flexible scope prototype will compared to standard of care scope used as standard of care.
  Arms: Patients evaluated using flexible nasopharyngoscope prototype device; Providers using flexible nasopharyngoscope prototype device

SUMMARY:
This study aims to develop and evaluate a low-cost, portable, flexible nasopharyngeal scope (FNS) used to assess head and neck cancers (HNC) in low resource settings. The FNS will be compared to an endoscope that is used as standard of care (SOC) in terms of ease of use, image quality, and perceived pain. The ultimate goal is to compare the ease of use between the FNS to what is used in SOC.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide signed and dated informed consent form
* Willing to comply with all study procedures and be available for the duration of the study
* Male or female, aged 18 or older
* Patients who clinical meet clinical criteria for SOC scope examination of the upper aerodigestive tract. This includes signs and symptoms such as dysphagia, nasal obstruction, neck mass, throat pain, and hoarseness.

Exclusion Criteria:

* Withdrawal of consent during the study duration
* Subjects who have complications from the SOC exam
* Anyone unable to under the SOC exam

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter Lee, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The providers who conducted the exams (n = 9) were not considered enrolled.
Groups:
- SOC Nasopharyngoscope Examination of the Upper Aerodigestive Tract: Participants who meet the clinical criteria to under a nasopharyngoscope examination were asked to have an exam with the study flexible nasopharyngoscope (FNS) after the routine scope exam done as part of their standard of care. They also completed a short survey about your experience with the investigational scope device compared to the routine scope exam.
Period: Exam With Standard Nasopharyngoscope
Arm/Group | SOC Nasopharyngoscope Examination of the Upper Aerodigestive Tract
Started | 53
Completed | 50
Not Completed | 3
Not completed — Study device not available | 2
Not completed — Withdrawal by Subject | 1
Period: Exam With Study Nasopharyngoscope
Arm/Group | SOC Nasopharyngoscope Examination of the Upper Aerodigestive Tract
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participants who completed the study are included.
Groups:
- SOC Nasopharyngoscope Examination of the Upper Aerodigestive Tract: Participants who meet the clinical criteria to under a nasopharyngoscope examination were asked to have an exam with the study flexible nasopharyngoscope (FNS) after the routine scope exam done as part of their standard of care. They also completed a short survey about their experience with the investigational scope device compared to the routine scope exam.
Arm/Group | SOC Nasopharyngoscope Examination of the Upper Aerodigestive Tract
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 35
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Participant Exams in Which Providers Reported the FNS (Flexible Nasopharyngoscope) is Easy to Use
Description: Measured using a 5 point scale, with 1=Very hard, 2=Harder, 3=Same, 4=Easier and 5=Very Easy.
Time Frame: up to 15 minutes
Population: Only applicable to the providers who conducted the exams.
Measure: Count of Units; unit: Participant exams
Units Other Than Participants: Participant exams
Arm/Group | Providers Using Flexible Nasopharyngoscope Prototype Device
Number analyzed (Participants) | 9
Number analyzed (Participant exams) | 50
Participant exams
  1=Very hard | 0
  2=Harder | 9
  3=Same | 33
  4=Easier | 6
  5=Very Easy | 2

2. Secondary Outcome: Image Quality of the Standard of Care (SOC) Scope as Measured on a 5-point Scale
Description: Measured using a 5 point scale where 1=poor, 2=fair, 3=good, 4=very good, and 5=excellent. Reported here is the number of participant exams in which providers scored the image quality of the SOC scope at each value.
Time Frame: Day 1
Population: Only applicable to the providers who conducted the exams.
Measure: Count of Units; unit: Participant exams
Units Other Than Participants: Participant exams
Arm/Group | Providers Using Flexible Nasopharyngoscope Prototype Device
Number analyzed (Participants) | 9
Number analyzed (Participant exams) | 50
Participant exams
  1=Poor | 0
  2=Fair | 0
  3=Good | 0
  4=Very Good | 14
  5=Excellent | 36

3. Secondary Outcome: Image Quality of the Flexible Scope as Measured on a 5-point Scale
Description: Measured using a 5 point scale where 1=poor, 2=fair, 3=good, 4=very good, and 5=excellent. Reported here is the number of participant exams in which providers scored the image quality of the flexible scope at each value.
Time Frame: Day 1
Population: Only applicable to the providers who conducted the exams.
Measure: Count of Units; unit: Participant exams
Units Other Than Participants: Participant exams
Arm/Group | Providers Using Flexible Nasopharyngoscope Prototype Device
Number analyzed (Participants) | 9
Number analyzed (Participant exams) | 50
Participant exams
  1=Poor | 0
  2=Fair | 0
  3=Good | 2
  4=Very Good | 13
  5=Excellent | 35

4. Secondary Outcome: Number of Patients Who Experienced an Adverse Event Following the Use of the Flexible Scope
Time Frame: Day 1
Population: Participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | SOC Nasopharyngoscope Examination of the Upper Aerodigestive Tract
Number analyzed (Participants) | 50
Participants | 0

5. Secondary Outcome: Number of Patients Who Experienced More, the Same, or Less Pain/Discomfort With the Flexible Scope Compared With the Standard of Care (SOC) Scope
Description: Comparison made using a 3 point scale where 1=much more, 2=about the same, and 3=much less.
Time Frame: Day 1
Population: Participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Providers Using Flexible Nasopharyngoscope Prototype Device
Number analyzed (Participants) | 50
Participants
  1=much more | 6
  2=about the same | 29
  3=much less | 15
Statistical Analysis 1: Comparison: Providers Using Flexible Nasopharyngoscope Prototype Device; Flexible scope compared with the SOC scope; Test type: Other; p = 0.04, Fisher Exact

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | SOC Nasopharyngoscope Examination of the Upper Aerodigestive Tract
All-Cause Mortality (participants affected / at risk) | 0/53
Serious Adverse Events (participants affected / at risk) | 0/53
Other Adverse Events (participants affected / at risk) | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-13): https://cdn.clinicaltrials.gov/large-docs/34/NCT04905134/Prot_SAP_001.pdf
  • Informed Consent Form (2023-09-13): https://cdn.clinicaltrials.gov/large-docs/34/NCT04905134/ICF_000.pdf